CLINICAL TRIAL: NCT05403463
Title: The Effect of Covid-19 on the Disease Course of Multiple Sclerosis
Brief Title: The Effect of Covid-19 on the Disease Course of Multiple Sclerosis :Belgian Lessons Learned From Rocky I to Rocky IV
Acronym: TofCoMS
Status: Completed | Type: Observational
Sponsor: Marie D'hooghe (Other)
Responsible Party: Sponsor-Investigator, Marie D'hooghe, neuroloog, National MS Center Melsbroek
Organization: National MS Center Melsbroek (Other)
Other Study IDs: TofComs
Record Dates: First submitted 2022-06-02; First posted 2022-06-03 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational cohort study. ToFCoMS: two years of follow-up of COVID-19 in MS.

DETAILED DESCRIPTION:
Methods The Nationaal Multiple Sclerose Centrum (NMSC) Melsbroek is a large highly-specialized center specifically focusing on neurological management, multidisciplinary care and rehabilitation in patients with MS. Since March 2020 (i.e., the onset of the pandemic in Belgium, and the first of five waves of spiking infection numbers thus far in our country), clinical data of patients followed at the center have been collected in a local database in case of COVID-19 diagnosis. The following items have been recorded: name, gender and date of COVID-19 diagnosis; age, Expanded Disability Status Scale score, MS duration, clinical subtype and DMT regimen at time of COVID-19 diagnosis; COVID-19 severity (method 1: categorized as ambulatory, hospitalized, death; method 2: categorized as asymptomatic, mild illness, moderate illness, severe illness, critical illness and death); vaccination status (categorized as non-vaccinated, fully vaccinated, fully vaccinated + booster) at time of COVID-19 diagnosis. On February 28, 2022, this database was locked and consisted of 234180 unique individual COVID-19 cases.

The NMSC Melsbroek features a second and more large database containing a broad variety of (para)clinical information gathered during routine follow-up, which includes regular testing of general disability with the EDSS, leg function/ambulation with the Timed 25-Foot Walk Test (T25FWT), hand function/dexterity using the 9-Hole Peg Test (9HPT) and cognition/information processing speed with the Symbol Digit Modalities Test (SDMT). For each of these parameters, the first two assessments before COVID-19 diagnosis (labelled T0 and T1, respectively; T1 is the closest to COVID-19 diagnosis), and the first thereafter (labelled T2), were retrieved for each COVID-19 subject. If clinical measurements were performed during an in-house stay for rehabilitation purposes, only those performed on admission were retained (thus not necessarily those the closest to the COVID-19 infection).

ELIGIBILITY:
Inclusion Criteria:

diagnosis of Multiple Sclerosis Covid 19 infection with PCR test

Exclusion Criteria:

other diagnosis than Multiple Sclerosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients with Covid 19 infection
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The investigators hereby aim to answer the question whether COVID-19 affects the progression of clinical disability in MS | 2 years
  The difference between the values measured at T-2 and T-1 (i.e., before COVID-19) will be compared, after adjustment for the time interval, with the difference between the respective values measured at T-1 and T1 (i.e., after COVID-19) for T25WT, 9HPT and SDMT. The investigators hereby aim to answer the question whether COVID-19 affects the progression of clinical disability in MS. Its effect on SDMT evolution has been defined as the primary endpoint of our study.

SECONDARY OUTCOMES:
vaccination status and progression MS | 2 years
  As secondary outcomes, the investigators want to explore whether (a) there is a relationship between COVID-19 severity and the evolution of clinical disability (i.e., differences between T-1 and T1), (b) vaccination status affects COVID-19 severity (in the total cohort as well as stratified according to DMT) and evolution of clinical disability (i.e., differences between T-1 and T1) and (c) DMT influences COVID-19 severity and evolution of clinical disability (i.e., differences between T-1 and T1).

CONTACTS AND LOCATIONS:
Locations (1):
- Nationaal MS center, Melsbroek, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
no IPD

REFERENCES:
- [Derived] Peeters G, Van Remoortel A, Nagels G, Van Schependom J, D'haeseleer M. Occurrence and Severity of Coronavirus Disease 2019 Are Associated With Clinical Disability Worsening in Patients With Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2023 Feb 17;10(3):e200089. doi: 10.1212/NXI.0000000000200089. Print 2023 May. PMID 36807080